CLINICAL TRIAL: NCT01387646
Title: Behavioral Intervention for Minority Adolescent Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jane Dimmitt Champion, University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01DA019180-01 (NIH); 1R01DA019180-01 (NIH)
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Sexually Transmitted Infection; Substance Use; Abuse; Pregnancy
Keywords: STI, abuse, substance use, unintended pregnancy
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Control Group (Other): Participants in the control arm will be interviewed at baseline, be given a targeted physical exam including a STI/HIV screen, pap smear and contraception counseling and will receive abuse and enhanced clinical counseling
  Interventions: Behavioral: Project IMAGE

INTERVENTIONS:
Behavioral: Project IMAGE — Participants in the intervention arm will be interviewed at baseline, given a targeted physical exam including a STI/HIV screen, pap smear and contraception counseling and enrolled in the intervention. The intervention will include 2 workshops, 5 support groups sessions and 2 individual counseling sessions. They will be interviewed and examined again after completing the intervention, to establish a post-intervention baseline.

SUMMARY:
The purpose of this Stage II clinical trial is to test the efficacy of a culturally sensitive, cognitive-behavioral intervention to reduce sexual risk behavior among minority adolescents for prevention of sexually transmitted infection (STI/HIV), unintended pregnancy and abuse by changing high-risk sexual behaviors, decreasing substance use and encouraging contraceptive use. Its primary goal is to expand risk-reduction interventions created in previous studies to further increase intervention efficacy for this particularly vulnerable, high-risk group. An adolescent intervention has been created and pilot tested in developmental studies. Results indicated reductions in substance use, risk behaviors, unintended pregnancy, STI and abuse without reports of adverse outcomes. Specific aims of the current study include: 1) To obtain a more in-depth understanding of configurations of psychosocial and situational factors associated with high-risk sexual behavior, substance use, STI/HIV and contraceptive use among abused minority adolescent women with STI; 2) To implement a controlled randomized trial of a cognitive behavioral risk-reduction intervention consisting of 2 small group sessions, 2 individual counseling and 3 support groups for this group; 3) To evaluate the effects of the adolescent intervention model versus enhanced counseling for this group on AIDS Risk Reduction Model (ARRM)-related constructs, high-risk sexual behavior, substance use, abuse recurrence, contraceptive use, unintended pregnancy and STI/HIV at 6 and 12 months follow-up. Participants will include a convenience sample of 600 Mexican-and African American adolescent women, aged 14-18 years with a history of sexual or physical abuse and current STI.

DETAILED DESCRIPTION:
African-and Mexican-American adolescent women with a current STI and history of abuse will be identified at public health and STI clinics within the San Antonio Metropolitan Health District system. Women who agree to participate and give informed consent will be randomized into the intervention or control arm. Women in the control arm will be interviewed at baseline, be given a targeted physical exam including a STI/HIV screen, pap smear and contraception counseling and will receive abuse and enhanced clinical counseling. Women in the intervention arm will be interviewed at baseline, given a targeted physical exam including a STI/HIV screen, pap smear and contraception counseling and enrolled in the intervention. Women in the intervention arm will be interviewed and examined again after completing the intervention, to establish a post-intervention baseline. All women in the study will be followed over one year, with follow-up interviews including an inquiry about any Adverse Events (AEs) or Serious Adverse Events (SAEs), and a targeted physical exams and contraception counseling at 6 and 12 months. During the study period, women will be encouraged to return to the study clinic for problem visits if they suspect they have been infected with a STI or require contraception or abuse counseling. All analyses of intervention effects will be performed on an intent-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 14-18 years, Mexican-or African-American female with a history of STI or abuse seeking health care through the San Antonio Metropolitan Health District.

Exclusion Criteria:

* No history of STI or abuse

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 562 (Actual)
Dates: Start 2004-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Sexually transmitted infection | 12 months
  Infection at 12 months with either chlamydia or gonorrhea

SECONDARY OUTCOMES:
Substance Use | 12 months
  Frequency and type of substance use
Experience of abuse | 12 months
  Type and frequency of experience of abuse
Unintended pregnancy | 12 months
  Frequency of unintended pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Jane D Champion, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- San Antonio Metropolitan Health District, San Antonio, Texas, United States

REFERENCES:
- [Derived] Collins JL, Owen DC, Champion JD. The Meaning of Weight: A Big Way of Life for Rural Mexican-American Adolescent Men and Caregivers. Public Health Nurs. 2016 Sep;33(5):421-9. doi: 10.1111/phn.12263. Epub 2016 Apr 14. PMID 27079291
- [Derived] Collins JL, Champion JD. Assessment of mobile device and SMS Use for Diet and Exercise Information Among Rural Mexican-American adolescents. J Pediatr Nurs. 2014 Nov-Dec;29(6):493-502. doi: 10.1016/j.pedn.2014.03.020. Epub 2014 Mar 15. PMID 24704179
- [Derived] Dimmitt Champion J, Harlin B, Collins JL. Sexual risk behavior and STI health literacy among ethnic minority adolescent women. Appl Nurs Res. 2013 Nov;26(4):204-9. doi: 10.1016/j.apnr.2013.06.003. Epub 2013 Jul 15. PMID 23867137